CLINICAL TRIAL: NCT06133972
Title: A Randomized, Double-blind, Placebo-controlled Extension Study to Assess the Long-term Safety and Tolerability of Ianalumab in Patients With Systemic Lupus Erythematosus (SIRIUS-SLE Extension)
Brief Title: Phase 3 Extension Study to Evaluate Long-term Safety of Ianalumab in Participants With Systemic Lupus Erythematosus (SIRIUS-SLE Extension).
Acronym: SIRIUS-SLE LTE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736F12301E1; 2023-505929-14-00 (Registry Identifier: EU CT NUMBER)
Expanded Access: NCT07244289 (Available)
Record Dates: First submitted 2023-10-02; First posted 2023-11-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; SLE; B cell depletion; SLEDAI-2K; BILAG-2004; SRI-4, ANA; ianalumab; VAY736
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — ianalumab

STUDY DESIGN:
Intervention Model Description: The trial is designed to evaluate long-term safety, tolerability and efficacy of two regimen of ianalumab versus placebo, given as monthly or quarterly subcutaneous (s.c.) injection
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ianalumab monthly (Experimental): Ianalumab s.c. monthly
  Interventions: Drug: Ianalumab
- Ianalumab quarterly (Experimental): Ianalumab s.c. quarterly
  Interventions: Drug: Ianalumab
- Placebo monthly (Placebo Comparator): Placebo s.c. monthly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo s.c. monthly
  Arms: Placebo monthly
Drug: Ianalumab — Ianalumab s.c. monthly Ianalumab s.c. quarterly
  Other Names: VAY736
  Arms: Ianalumab monthly; Ianalumab quarterly

SUMMARY:
The purpose of this study is to evaluate long-term safety and tolerability of ianalumab in participants with systemic lupus erythematosus who have previously completed the treatment period in one of the two SIRIUS-SLE core studies (CVAY736F12301 or CVAY736F12302).

DETAILED DESCRIPTION:
The purpose of this extension study is to evaluate long-term safety and tolerability of ianalumab administered s.c. monthly or quarterly, compared to monthly placebo, in adolescent and adult participants with anti-nuclear antibody (ANA)-positive systemic lupus erythematosus of moderate-to-severe disease activity, who have completed either CVAY736F12301 (SIRIUS-SLE 1) or CVAY736F12302 (SIRIUS-SLE 2) core studies.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent prior to participation in the extension study. Parent or legal guardian's signed informed consent and child's assent, if appropriate, are required before any assessment is performed for participants <18 years of age. Of note, if the participant reaches age of consent (age as per local law) during the study, they will also need to sign the corresponding study Informed Consent Form (ICF) at the next study visit.
* Participants must have participated in either one of the two SIRIUS-SLE core studies, CVAY736F12301 or CVAY736F12302, and have completed the treatment period through Week 60 without treatment discontinuation.
* In the judgement of the investigator, participants must be expected to clinically benefit from continued study treatment.

Key Exclusion Criteria:

* Use of prohibited therapies.
* Active viral, bacterial or other infections requiring intravenous or intramuscular treatment for clinically significant infection which in the opinion of the investigator will place the participant at risk for participation.
* Plans for administration of live vaccines during the study period.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, refusing or unable to use highly effective methods of contraception while on study treatment and for 6 months after stopping of study drug (or longer if required by concomitant medications).
* United States (and other countries, if locally required): sexually active males, unless they agree to use barrier protection during intercourse with women of child-bearing potential while taking study treatment.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2030-04-19 (Estimated); Study Completion 2032-04-16 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-emergent Adverse events/Serious Adverse events | through study completion, up to approximately 91 months
  Assessment of long-term safety and tolerability of ianalumab

SECONDARY OUTCOMES:
Proportion of participants who achieved Systemic Lupus Erythematosus Responder Index -4 (SRI-4) response | up to Week 216
  SRI-4 response is defined as:
  * Systemic Lupus Erythematosus Disease Activity Index - 2000 (SLEDAI-2K) reduction from baseline of ≥ 4 points
  * No British Isles Lupus Assessment Group-2004 (BILAG-2004) worsening, defined as ≥ 1 new A or ≥ 2 new B items compared to baseline
  * No worsening in Physician Global Assessment of Disease Activity (PhGA), defined as an increase of ≥ 0.3 from baseline on a 0 to 3 visual analog scale
Change in Systemic Lupus International Collaborating Clinics/American College of Rheumatology (SLICC/ACR) Damage Index | up to Week 216
  SLICC/ACR Damage Index is a measure of cumulative damage due to SLE
Average daily dose of oral corticosteroids administered | up to Week 216
  Evaluating the effect of ianalumab on corticosteroids intake
Annualized BILAG moderate or severe flare rate | up to Week 216
  Annualized BILAG moderate or severe flare rate where moderate BILAG flare is defined as 2 or more new BILAG-2004 B items, and severe BILAG flare is defined as 1 or more new BILAG-2004 A items, compared to the previous visit

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (104):
- United States (18):
  - Pinnacle Research Group Llc, Anniston, Alabama
  - Providence Medical Center, Burbank, California
  - Advanced Medical Research, La Palma, California
  - Millennium Clinical Trials, Westlake Village, California
  - University of Colorado Denver, Aurora, Colorado
  - Clinical Res Of W Florida, Clearwater, Florida
  - GNP Research, Cooper City, Florida
  - IRIS Research and Development, Plantation, Florida
  - Robert A Hozman MD SC, Skokie, Illinois
  - Willow Rheumatology Wellness, Willowbrook, Illinois
  - Accurate Clinical Research, Lake Charles, Louisiana
  - Henry Ford Health, Detroit, Michigan
  - Ahmed Arif Medical Research Center, Grand Blanc, Michigan
  - Paramount Med Rsrch and Consult LLC, Middleburg Heights, Ohio
  - West Tennessee Research Institute, Jackson, Tennessee
  - Shelby Research LLC, Memphis, Tennessee
  - Novel Research LLC, Bellaire, Texas
  - Accurate Clinical Research, League City, Texas
- Argentina (4):
  - Novartis Investigative Site, San Miguel, Buenos Aires
  - Novartis Investigative Site, San Miguel, Tucumán Province
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, San Miguel de Tucumán
- Novartis Investigative Site, Maroochydore, Queensland, Australia
- Brazil (6):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Salvador
- Bulgaria (2):
  - Novartis Investigative Site, Plovdiv, Bulgaria
  - Novartis Investigative Site, Sofia
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Rimouski, Quebec
- Chile (3):
  - Novartis Investigative Site, Valdivia, Los Ríos Region
  - Novartis Investigative Site, Santiago, RM
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
- China (12):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Pingxiang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Linyi, Shandong
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Ningbo, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Colombia (5):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Chía, Cundinamarca
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Bogotá
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Uherské Hradiště
- France (3):
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Novartis Investigative Site, Leipzig, Saxony, Germany
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City, Departamento de Guatemala
  - Novartis Investigative Site, Guatemala City
- Hungary (2):
  - Novartis Investigative Site, Székesfehérvár, Fejér
  - Novartis Investigative Site, Gyula
- India (5):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Kozhikode, Kerala
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, New Delhi
- Israel (2):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
- Novartis Investigative Site, Torino, TO, Italy
- Japan (3):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Chuo Ku, Tokyo
- Novartis Investigative Site, Ipoh, Perak, Malaysia
- Mexico (6):
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Morelia, Michoacán
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, México
- Poland (4):
  - Novartis Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Bytom
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, Braga, Portugal
- Romania (3):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
- Novartis Investigative Site, Cape Town, Western Cape, South Africa
- South Korea (2):
  - Novartis Investigative Site, Gwangju Gwangyeoksi, Gwangju
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, San Sebastian Reyes, Madrid
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com